CLINICAL TRIAL: NCT05174091
Title: A Comparıson of Functıonal Movemenet Screen, Physıcal Capacıty, Core Endurance, and Spınal Mobılıty in People Wıth and Wıthout Non-Specıfıc Low Back Paın
Brief Title: A Comparıson of in People Wıth and Wıthout Non-Specıfıc Low Back Paın
Status: Completed | Type: Observational
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Fatih ÖZYURT, Principal Investigator, University of Beykent
Other Study IDs: 15212021
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Low Back Pain
Keywords: Functional; Movement; Screen; Core; Endurance; Physical capacity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Non- Spesific Low Back Pain: FMS, Spinal mobility, Core Endurance, Physical Capacity.
  Interventions: Other: Functional Movement Screen, Spinal Mouse, Core Endurance, Funcitonal Capacity
- Without Non- Spesific Low Back Pain: FMS, Spinal mobility, Core Endurance, Physical Capacity.
  Interventions: Other: Functional Movement Screen, Spinal Mouse, Core Endurance, Funcitonal Capacity

INTERVENTIONS:
Other: Functional Movement Screen, Spinal Mouse, Core Endurance, Funcitonal Capacity — Due to the difficulties in the diagnosis and treatment of NSLBP, it has been causing many problems such as limitation of activation, socioeconomic burden, and biopsychosocial factors for years. It is thought that the effectiveness of treatment will increase if the needs and problems of individuals with NSLBP are clearly revealed beforehand. Although there are studies on core endurance and physical capacities in individuals with NSLBP in the literature, the number of studies examining functional movement analysis and spinal mobility in individuals with NSLBP is very few. Therefore, aim of this research is to compare functional movement analysis, physical capacity, core endurance, and spinal mobility in individuals with and without NSLBP. With the results we will reveal, we aim to contribute to the evaluation and treatment of patients with NSLBP. Thus, the negative effects of this pathology, which causes serious labor and financial losses, can be minimized.

SUMMARY:
Non-Specific Low Back Pain (NSLBP), which constitutes approximately 90-95% of low back pain, is low back pain that cannot be defined by specific pathologies such as infection, tumor, osteoporosis, fracture, radicular symptoms or inflammatory diseases. NSLBP creates many health problems due to uncertainties in both its diagnosis and treatment. Due to the health problems and decreased functional activities of the individual, it creates a socioeconomic burden on both the individual and the country. NSLBP ranks 6th in the distribution of the economic burden caused by diseases to developed and developing societies. It is difficult to calculate how much burden it puts on the country's economy both directly (health institutions) and indirectly (loss of working days). However, in 1996 in the United States (USA), the economic burden of NSLBP patients is estimated to be between 18.5 and 28.2 million.

DETAILED DESCRIPTION:
Non-Specific Low Back Pain (NSLBP), which constitutes approximately 90-95% of low back pain, is low back pain that cannot be defined by specific pathologies such as infection, tumor, osteoporosis, fracture, radicular symptoms or inflammatory diseases. NSLBP creates many health problems due to uncertainties in both its diagnosis and treatment. Due to the health problems and decreased functional activities of the individual, it creates a socioeconomic burden on both the individual and the country. NSLBP ranks 6th in the distribution of the economic burden caused by diseases to developed and developing societies. It is difficult to calculate how much burden it puts on the country's economy both directly (health institutions) and indirectly (loss of working days). However, in 1996 in the United States (USA), the economic burden of NSLBP patients is estimated to be between 18.5 and 28.2 million.

Although the age of first appearance of NSLBP is in the middle of the second decade and the beginning of the third decade, its prevalence increases until the middle of the sixth decade. NSLBP, which is more common in women aged 40-69 years, is more common in high-income countries. Due to the complex nature of the etiology of NSLBP, it is very difficult to define the risk factors. However, there may be many risk factors such as age, race, gender, muscle strength, body mass index, smoking, spine mobility. Since the underlying cause is not clear, there is currently no suitable evaluation and treatment method. For this, the patient's muscle strength, endurance, range of motion, physical capacity and functional movement analysis should be evaluated and interpreted.

ELIGIBILITY:
Inclusion Criteria for the NSLBP:

* Being between the ages of 18-65,
* getting more than 24 points in the minimental test,
* having pain between the last rib and inferior gluteal region,
* being diagnosed with NSLBP, presence of low back pain for more than 3 months, -volunteering to participate in the study.

Inclusion criteria for the Without NSLBP group;

* Being between the ages of 18-65,
* getting over 24 points in the minimental test,
* not having low back pain in the last 3 months,
* volunteering to participate in the study were determined.

Exclusion Criteria:

* uncontrollable hypertension and heart disease,
* uncontrollable neurological and metabolic disease,
* trauma history in the last 6 months,
* serious musculoskeletal problem and other pathology that may adversely affect balance,
* severe mental involvement, lower extremity amputation,
* presence of nerve pressure, non-voluntary

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18-65, • having pain between the last rib and inferior gluteal region more than 3 months
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screening (FMS) (Functional Movement Patterns) | 1 day
  FMS will be used to evaluate the quality of 7 functional movement patterns with the goal of identifying movement limitations and asymmetries. The FMS consists of 7 individual test items including the deep squat, in-line lunge, hurdle step, shoulder flexibility, push-up, straight leg raise, and rotary trunk stability assessment. Each of these 7 test items is graded on a scale of 0-3; thus, the lowest and highest possible overall FMS scores are 0 and 21, respectively.
Spinal Mobility | 1 day
  Spinal mobility will be measured with a computer-assisted portable electromechanical device (the Spinal Mouse System, Idiag, Fejraltorf, Switzerland). Measurements will be made with the participant's back naked. Spinous processes between C7 and S3 of the individual will be marked before spinal mouse measurement is made. The C7 spinous process is located between the two rounds of the spinal mouse. It will go down to the S3 vertebra with a speed of 6.7 cm/sec, which measures without disturbing the patient's position. Then, the same measurements will be made between the C7 spinous process and the S3 spinous process while the person is in the position of maximum flexion, extension and right-left lateral flexion.

SECONDARY OUTCOMES:
Oswetry Disability Index | 1 day.
  Patients with NSBA may have limitations in activities of daily living. In this study, the disability level of low back pain will be measured with the Oswestry Low Back Pain Disability Questionnaire (ODI). ODI evaluates the person's disability with 10 questions. Each of the titles of pain intensity, personal care activities, lifting, walking, sitting, standing, sleep, sexual life, social life and travel activities are scored between 0-5. The maximum score received in the survey is 100. High scores are associated with higher disability from low back pain.
Functional Reach Test | 1 day.
  The Functional Reach Test is a test used to assess balance. Participants will be asked to stand with their feet shoulder-width apart. There will be a measuring stick attached to the wall at the participant's shoulder level. The participant will be asked to bring the third metacarpophalangeal joint to the starting point of the measuring stick, without touching the wall, with the shoulder joint 90 degrees flexed, elbow in full extension, and hand in the form of a fist. After the physiotherapist who made the assessment marks the starting point, the participant will be asked to reach the maximum distance they can reach without taking a step. The endpoint will be saved at the endpoint. The distance between the start and end point in cm will be measured and recorded. The test will be repeated 3 times and the best score will be recorded
Two Minutes Step Test | 1 day.
  The Two Minute Step Test is a test used to assess a participant's aerobic capacity. It is preferred in the clinic because it can be done in a shorter time than the Six Minute Walk Test, it is safe and does not require expensive equipment. The middle distance between the participant's iliac crest and patella will be marked on the wall. After the test starts, the participant will be asked to take a step on the spot by extending the knee up to the marked line. The number of times the participant brought his right knee up to the line for two minutes will be recorded as the score. The test will be administered once.
Time Up and Go Test | 1 day.
  The Timed Up and Go Test is a test used to evaluate dynamic balance and mobility. This test includes motor tasks such as getting up, walking straight, turning and sitting. Participants will be asked to get up from their seat, turn from the place 3 meters ahead and return to the chair they started from again. The total test time will be recorded in seconds. The test will be repeated 2 times in total and the average of the data obtained will be recorded.
The Trunk Flexor Endurance Test | 1 day
  The Trunk Flexor Endurance Test is a test that evaluates the endurance of the rectus abdominus muscle. In this test, the participant reclines with his arms crossed at chest level, hips and knees positioned at 90 degrees of flexion, while the top of the bed is at 60 degrees. With the start of the test, the back of the participant who is supported by the bed stays up 10 cm from the bed. The test is terminated when the participant's back touches the bed. The elapsed time is recorded in seconds.
The Trunk Extensor Endurance Test | 1 day
  The Trunk Extensor Muscles Endurance Test is a test used to evaluate the endurance of the muscles in the back of the back. In the prone position, the lower extremity is supported by a belt while the participant is suspended out of the bed at the level of the anterior superior spina illiaca. Before the test starts, the participant carries his weight with the help of a chair, while the chair is taken at the start of the test and the arms are extended parallel to the ground beside the torso. The test is terminated when the participant's body becomes uneven and the elapsed time is recorded in seconds
Trunk Lateral Muscle Endurance Test | 1 day.
  In the Trunk Lateral Muscle Endurance test, it is a test used to evaluate the endurance of the internal and external oblique muscles on the lateral side of the abdominal region. The participant places one elbow under his shoulder at 90 degrees of flexion. While the legs are in the extension position in line with the body, the top foot is placed under the bottom foot. The upper hand is placed on the opposite shoulder. The time spent by the participant in this position will be recorded in seconds and repeated for the other party.
Numeric Pain Rating Scale | 1 day.
  The pain intensity of the patients will be measured with the numerical pain intensity scale. On the numerical pain intensity scale, the patient will be asked to give a value between 0 and 10 for his pain. The size of the score indicates that the severity of pain is high.
Sociodemographic Information | 1 day
  Age (year), height (cm), body weight (kg), body mass index (kg/m2), marital status, duration of pain (months), severity of pain (0-10), location of pain (right) , left, middle), dominant upper extremity (writing hand), occupation, whether the occupation requires movement, education level, smoking and alcohol use, exercise habits, medications used, background, family history and accompanying diseases will be questioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Beykent University, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmadi H, Adib H, Selk-Ghaffari M, Shafizad M, Moradi S, Madani Z, Partovi G, Mahmoodi A. Comparison of the effects of the Feldenkrais method versus core stability exercise in the management of chronic low back pain: a randomised control trial. Clin Rehabil. 2020 Dec;34(12):1449-1457. doi: 10.1177/0269215520947069. Epub 2020 Jul 29. PMID 32723088
- [Background] Kellis E, Adamou G, Tzilios G, Emmanouilidou M. Reliability of spinal range of motion in healthy boys using a skin-surface device. J Manipulative Physiol Ther. 2008 Oct;31(8):570-6. doi: 10.1016/j.jmpt.2008.09.001. PMID 18984239
- [Background] Vachalathiti R, Sakulsriprasert P, Kingcha P. Decreased Functional Capacity in Individuals with Chronic Non-Specific Low Back Pain: A Cross-Sectional Comparative Study. J Pain Res. 2020 Aug 5;13:1979-1986. doi: 10.2147/JPR.S260875. eCollection 2020. PMID 32801853
- [Background] Cook G, Burton L, Hoogenboom B. Pre-participation screening: the use of fundamental movements as an assessment of function - part 1. N Am J Sports Phys Ther. 2006 May;1(2):62-72. PMID 21522216
- See also: This artickle linked to our research — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2953313/